CLINICAL TRIAL: NCT00567281
Title: Bilateral rTMS Clinical Trial for Persistent Auditory Hallucinations Original Study
Brief Title: Bilateral Repetitive Transcranial Magnetic Stimulation for Auditory Hallucinations Original Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Device Feasibility
Other Study IDs: 0409027023_a; R01MH073673-02 (NIH); NARSAD; 2R01MH067073 (NIH)
Record Dates: First submitted 2007-12-03; First posted 2007-12-04 (Estimated); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Schizophrenia
Keywords: Schizoaffective disorder; Auditory Hallucinations; Voices; Repetitive Transcranial Magnetic Stimulation; rTMS; Wernicke's Area; Middle Temporal Cortex; Persistent Auditory Hallucinations; Previously Participated in "Parent" rTMS Protocol
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Hallucinations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Active bilateral rTMS to left/right Wernicke's area and opposite side middle temporal gyrus
  Interventions: Device: Magstim Rapid 2 system triggering Magstim Super Rapid system
- 2 (Active Comparator): Active rTMS to left/right Wernicke's region plus sham rTMS to opposite hemisphere middle temporal cortex
  Interventions: Device: Magstim Rapid-2 system triggering Magstim Super Rapid system

INTERVENTIONS:
Device: Magstim Rapid 2 system triggering Magstim Super Rapid system — Week 1 treatment includes rTMS for 5 sessions to either to left or right Wernicke's area (BA22) synchronous with rTMS to opposite hemisphere middle temporal cortex (BA21). Week 2 treatment includes rTMS given for 5 sessions with positions reversed (e.g., if Wernicke's stimulation was on the left during Week 1, position of rTMS will switch to the right side during Week 2 and vice-versa). As in Week 1, active rTMS will also be given synchronously to the opposite hemisphere middle temporal cortex. Weeks 3 and 4 include 10 stimulation sessions to the configuration of sites producing greater improvement in comparing results of Week 1 and Week 2. rTMS for each stimulation session will be given at 1-Hertz (once per second) for 16 minutes without interruption.
  Arms: 1
Device: Magstim Rapid-2 system triggering Magstim Super Rapid system — Week 1 includes repetitive rTMS for 5 sessions to either to left or right Wernicke's area (BA22) synchronous with sham rTMS to opposite hemisphere middle temporal cortex (BA21). Week 2 includes rTMS given for 5 sessions with positions reversed (e.g., if Wernicke's stimulation was on the left during Week 1, position of rTMS will switch to the right side during Week 2 and vice-versa). As in Week 1, sham rTMS will also be given synchronously to the opposite hemisphere middle temporal cortex. Weeks 3 and 4 include 10 stimulation sessions to the configuration of sites producing greater improvement in comparing results of Week 1 and Week 2. rTMS for each stimulation session will be given at 1-Hertz (once per second) for 16 minutes without interruption.
  Arms: 2

SUMMARY:
This trial is designed to determine if administering repetitive transcranial magnetic stimulation (rTMS) simultaneously to two sites in the temporal lobes, one on the left and one on the right, produces greater improvements in "voices" and other symptoms of schizophrenia compared to rTMS given to just one site in the temporal lobes.

DETAILED DESCRIPTION:
This study is an extension of an ongoing clinical trial (ClinicalTrials.gov identifier NCT 00308997) that was initiated in 2006. The primary objective of the ongoing clinical trial (hereafter called the "parent trial") is to determine efficacy of rTMS in curbing auditory hallucinations when delivered to a part of the left temporal lobe called Wernicke's area and a corresponding region in the right temporal lobe. The parent trial appears to show robust effects for active rTMS compared to effects of sham stimulation. However, observed responses following active rTMS have often been incomplete. Moreover, in some cases there has been a subsequent return of symptoms 1 to 6 months after the trial ended.

We consequently have initiated a trial where patients who have participated in the parent trial and demonstrated an incomplete response or a subsequent return of symptoms may return to receive additional active rTMS. We hypothesize that efficacy of suppressive rTMS will be enhanced if directed simultaneously to right/left Wernicke's area (the site used in the parent trial) as well as to a second site located in the opposite middle temporal cortex. Roughly half of subjects in the re-enrollment will be randomized to receive active rTMS to right/left Wernicke's area plus active rTMS to opposite hemisphere middle temporal region, while half of subjects will be randomized to receive active rTMS to right/left Wernicke's area plus sham rTMS to opposite hemisphere middle temporal region. The position of the middle temporal regions will be determined by two recently completed brain imaging studies of auditory hallucinations suggesting that activation in these sites triggers auditory hallucinations. The two-position design will allow us to determine if active rTMS delivered to the middle temporal cortex is superior in amplifying efficacy of active rTMS targeting Wernicke's area and in reducing auditory hallucinations to sham stimulation to the same site. The re-enrollment protocol will utilize two rTMS devices simultaneously where one directly triggers the other.

This study record has been amended to remove a third arm that was added in 2012. The third arm described was not actually a comparative arm, but rather an added objective with a different study population. Dr. Ralph Hoffman unexpectedly passed away while this study was being conducted. This study has been submitted as a separate study (NCT04548622) where the summarized study results of the terminated study will be presented.

ELIGIBILITY:
Inclusion Criteria:

* Previously enrolled in our "parent" rTMS trial with passage of at least six months since last received active rTMS

Exclusion Criteria:

* Active substance abuse or alcohol abuse
* Pregnancy
* Dose or type of psychiatric medication changed within the 4 weeks prior to study entry
* Recent head trauma, seizures, or significant unstable medical condition

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2007-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Hallucination change score | Measured at every week over a total 4 weeks
Clinical Global Improvement Scale | Measured at every week over a total of 4 weeks
Frequency subscale of Auditory Hallucinations Rating Scale | Measured at baseline and every week over a total of 4 weeks

SECONDARY OUTCOMES:
Summed scores of Auditory Hallucination Rating Scale | Measured at baseline and every week over a total of 4 weeks
PANSS composite positive symptoms scale | Measured at baseline and every week over a total of 4 weeks
PANSS composite negative symptom scale | Measured at baseline and every week over a total of 4 weeks
PANSS total score | Measured at baseline and every week over a total of 4 weeks
California Verbal Learning Test (CVLT) | Measured at baseline and every week over a total of 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Hoffman, MD, Principal Investigator — Yale University
Locations (1):
- Department of Psychiatry, Yale School of Medicine, New Haven, Connecticut, United States

REFERENCES:
- [Background] Hoffman RE, Gueorguieva R, Hawkins KA, Varanko M, Boutros NN, Wu YT, Carroll K, Krystal JH. Temporoparietal transcranial magnetic stimulation for auditory hallucinations: safety, efficacy and moderators in a fifty patient sample. Biol Psychiatry. 2005 Jul 15;58(2):97-104. doi: 10.1016/j.biopsych.2005.03.041. PMID 15936729
- [Background] Hoffman RE, Boutros NN, Hu S, Berman RM, Krystal JH, Charney DS. Transcranial magnetic stimulation and auditory hallucinations in schizophrenia. Lancet. 2000 Mar 25;355(9209):1073-5. doi: 10.1016/S0140-6736(00)02043-2. PMID 10744097
- [Background] Hoffman RE, Hampson M, Wu K, Anderson AW, Gore JC, Buchanan RJ, Constable RT, Hawkins KA, Sahay N, Krystal JH. Probing the pathophysiology of auditory/verbal hallucinations by combining functional magnetic resonance imaging and transcranial magnetic stimulation. Cereb Cortex. 2007 Nov;17(11):2733-43. doi: 10.1093/cercor/bhl183. Epub 2007 Feb 13. PMID 17298962
- [Background] Hoffman RE, Anderson AW, Varanko M, Gore JC, Hampson M. Time course of regional brain activation associated with onset of auditory/verbal hallucinations. Br J Psychiatry. 2008 Nov;193(5):424-5. doi: 10.1192/bjp.bp.107.040501. PMID 18978327
- See also: Click here for a description of rTMS trials of auditory hallucinations at Yale — http://www.med.yale.edu/psych/clinics/rTMS.html